CLINICAL TRIAL: NCT04490421
Title: A Single-arm, Prospective Study of Camrelizumab Combined With Apatinib, Etoposide and Cisplatin in First-line Treatment of Extensive Small-cell Lung Cancer.
Brief Title: Camrelizumab Combined With Apatinib, Etoposide and Cisplatin Treat Small-cell Lung Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-FJ-SCLC-II-005
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-07

CONDITIONS: Lung Neoplasm; Small Cell Lung Cancer; PD-1 Inhibitors
Keywords: Small-cell lung cancer, immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — apatinib; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Experimental:Camrelizumab combined with Apatinib, Etoposide and Cisplatin
  Interventions: Drug: Camrelizumab combined with Apatinib, Etoposide and Cisplatin

INTERVENTIONS:
Drug: Camrelizumab combined with Apatinib, Etoposide and Cisplatin — Camrelizumab combined with Apatinib, Etoposide and Cisplatin

SUMMARY:
Small cell lung cancer is a highly malignant tumor, and its first-line treatment has not broken through platinum-containing dual-drug chemotherapy in the past 30 years. Because small cell lung cancer has the characteristics of easy resistance after first-line chemotherapy, increased difficulty in treatment after resistance, and poor efficacy of second-line treatment, how to formulate a plan that can control tumor progression to the greatest extent has become a hot issue in recent research. Recently, immunotherapy and targeted therapy have made breakthrough progress in small cell lung cancer, but its efficacy still needs to be further improved. As immune combined chemotherapy combined with targeted therapy first achieved good results in other tumors, this study aims to explore a longer disease-free survival time and higher overall survival rate of patients with small cell lung cancer through immunotherapy combined with targeted therapy combined with chemotherapy. Program to bring new hope to patients. At the same time, this study will evaluate the safety of the program, explore the prognostic indicators that may exist in the treatment, and provide new inspiration for subsequent patient selection.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and ≤75 years old, regardless of gender;
* Extensive-stage small cell lung cancer confirmed by histology or pathology;
* According to the RECIST V1.1 standard, there is at least one measurable lesion;
* Patients who have not previously been treated for small cell lung cancer (immune, targeted, chemotherapy, etc.);
* Eastern Cooperative Oncology Group's physical status score (ECOG PS) 0~1;
* Expected survival period ≥ 3 months;
* Women of childbearing age must undergo a serum pregnancy study within 2 weeks before the first medication, and the result is negative. Female subjects of childbearing age and male subjects whose partners are women of childbearing age must contraception during the study and within 180 days after the last administration of the study drug;
* The laboratory examination values of patients before medication must meet the following standards:

Blood routine: WBC≥3.0 × 109/L；ANC≥1.5 × 109/L；PLT≥100× 109/L；HGB≥9.0 g/dL; Liver function: TBIL≤1.5 × ULN, AST≤2.5 × ULN, ALT≤2.5 × ULN (for subjects with liver metastases, AST≤5×ULN, ALT≤5 × ULN) Renal function: Cr≤1.5 × ULN or CrCl ≥50 mL/min Coagulation function: INR≤1.5, APTT≤1.5 ×ULN

* The subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

* Active, known or suspected autoimmune diseases;
* Prior T cell co-stimulation or immunocheckpoint therapy, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other T-cell-targeted drugs;
* Interstitial lung disease, drug-induced pneumonia, radioactive pneumonia requiring steroid treatment or active pneumonia with clinical symptoms or severe pulmonary dysfunction;
* A past or present history of cancer other than SCLC, except for non-melanoma skin cancer, cervical cancer in situ, or other cancers that have received curative treatment and have not shown signs of recurrence for at least 5 years;
* Standard treatment for uncontrolled hypertension (blood pressure < 150/90 mmHg)
* Hereditary bleeding tendency or coagulation dysfunction. There were clinically significant bleeding symptoms or definite bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, and fecal occult blood ++ or above at baseline;
* Patients with definite or suspected brain metastases. Patients with a history of brain metastases must have completed treatment and no longer require corticosteroid therapy to be enrolled; For asymptomatic patients with no more than 3 lesions and a single brain transfer less than 10mm, the researcher judged whether they were included or not.
* Clinical symptoms or diseases of the heart that are not well controlled, such as :heart failure of NYHA2 or above; unstable angina pectoris; myocardial infarction within 24 weeks; clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
* The presence of clinically uncontrollable third interstitial effusion (such as pleural effusion/pericardial effusion, patients who do not need drainage or have no significant increase of effusion after 3 days of drainage can be enrolled);
* Subjects with a history of severe infection within 4 weeks prior to the first administration, including but not limited to infectious complications requiring hospitalization, bacteremia, severe pneumonia, etc. Subjects with any active infection were excluded. Lymphatic spread of lung cancer was not excluded.
* Imaging (CT or MRI) shows that the tumor invades the great vessels or the researchers judge that the tumor is likely to invade the important vessels and cause fatal hemorrhage during the follow-up study;
* A history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
* Active hepatitis B (defined as hepatitis B virus surface antigen [HBsAg] test positive and hbV-DNA test value higher than the upper limit of normal value in the laboratory of the research center) or Hepatitis C (defined as hepatitis C virus surface antibody [HCsAb] test positive and HCV-RNA positive);
* Subjects requiring systematic treatment with corticosteroids (>10 mg/ day prednisone or its equivalent) or other immunosuppressive agents within 14 days of the first administration. Adrenal hormone replacement therapy with inhaled or topical corticosteroids and > 10 mg/ day dose of prednisone in the absence of active autoimmune disease;
* Patients who received oral or intravenous antibiotics within 14 days before treatment;
* The patient has an allergic reaction to the experimental drug;
* Subjects who have received or will receive live vaccine within 30 days before the first medication;
* As determined by the researcher, the subjects have other factors that may lead to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival rate(1-year OS%) | up to 1-year
  1-year OS%, determined by RECIST V1.1 standard which means proportion of outcome events occurring within one year from the start of the trial

SECONDARY OUTCOMES:
progression-free survival(PFS) | up to approximately 4-6 months
  PFS, determined by RECIST V1.1 standard which means the time from the beginning of the organised clinical trial to the onset of tumors (in any aspect) or death due to any reason
overall survival(OS) | up to approximately 18 months
  OS, determined by RECIST V1.1 standard which means the time from randomization of patients in clinical trials to death due to any cause.
Objective Response Rate(ORR) | up to 1-year
  ORR, determined by RECIST V1.1 standard which refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time
disease control rate(DCR) | up to 1-year
  DCR, determined by RECIST V1.1 standard which refers to proportion of patients whose tumors have shrunk or stabilized for a certain period of time

CONTACTS AND LOCATIONS:
Overall Officials: Xiong Chen, Study Chair — The 900th Hospital of Joint Logistic Support Force
Locations (1):
- The 900th Hospital of Joint Logistic Support Force, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided